CLINICAL TRIAL: NCT02231008
Title: A Double-blind, Randomized, Two-period Crossover Study Evaluating the Effects of Tasimelteon vs. Placebo on Sleep Disturbances of Individuals With Smith-Magenis Syndrome (SMS)
Brief Title: Evaluating the Effects of Tasimelteon vs Placebo on Sleep Disturbances in SMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VP-VEC-162-2401
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Smith-Magenis Syndrome; Circadian
Keywords: SMS
MeSH Terms: conditions — Smith-Magenis Syndrome | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tasimelteon (Experimental): Single dose oral capsule or equivalent age-appropriate oral formulation, daily dosage
  Interventions: Drug: tasimelteon
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tasimelteon
  Arms: Tasimelteon
Drug: placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate tasimelteon vs. placebo on sleep disturbances of individuals with Smith-Magenis Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed clinical diagnosis of SMS
2. Informed consent from the patient or the legal guardian
3. Male or female between the ages of 3- 65 years of age
4. Recent history of sleep disturbances
5. Have an appointed care-giver complete the required outpatient assessments
6. Willing and able to comply with study requirements and restrictions

Exclusion Criteria:

1. Unable to dose daily with medication
2. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever was longer) of screening
3. Any other sound medical reason as determined by the clinical investigator

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of tasimelteon administered daily compared to placebo, as measured by improvement in sleep parameters | 9 Weeks

SECONDARY OUTCOMES:
Safety and tolerability as measured by spontaneous reporting of adverse events (AEs). | up to 137 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Santa Monica, California
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Houston, Texas